CLINICAL TRIAL: NCT06037148
Title: A Phase I Dose Escalation Trial to Investigate the Safety, Tolerability, and Explorative Efficacy, Following Environmental Allergen Exposure in a Chamber, of DM-101PX in Participants With Birch Pollen Allergy
Brief Title: Study to Evaluate Safety, Tolerability and Explorative Efficacy of DM-101PX in Birch Pollen Allergic Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Desentum Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: DM-101-C-002
Record Dates: First submitted 2023-09-06; First posted 2023-09-14 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Birch Pollen Allergy

STUDY DESIGN:
Intervention Model Description: 3 sequential dose cohorts with ascending DM-101PX doses. In each cohort two treatment arms: placebo and active drug
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DM-101PX low dose (Experimental): 10 subcutaneous doses starting from 0.05 ug of which first 8 doses are ascending. Thereafter the 8th dose is repeated twice. First 9 doses are administered at 1 week interval, and the 10th dose is administered 2 weeks after the 9th dose.
  Interventions: Biological: DM-101PX
- Placebo (Placebo Comparator): 10 subcutaneous doses.First 9 doses are administered at 1 week interval, and the 10th dose is administered 2 weeks after the 9th dose.
  Interventions: Biological: Placebo to Match DM-101PX
- DM-101PX middle dose (Experimental): 10 subcutaneous doses starting from 0.1 ug of which first 8 doses are ascending. Thereafter the 8th dose is repeated twice. First 9 doses are administered at 1 week interval, and the 10th dose is administered 2 weeks after the 9th dose.
  Interventions: Biological: DM-101PX
- DM-101PX high dose (Experimental): 10 subcutaneous doses starting from 0.2 ug of which first 8 doses are ascending. Thereafter the 8th dose is repeated twice. First 9 doses are administered at 1 week interval, and the 10th dose is administered 2 weeks after the 9th dose.
  Interventions: Biological: DM-101PX

INTERVENTIONS:
Biological: DM-101PX — subcutaneous injection of DM-101PX
  Arms: DM-101PX high dose; DM-101PX low dose; DM-101PX middle dose
Biological: Placebo to Match DM-101PX — Placebo to match DM-101PX administered subcutaneously
  Arms: Placebo

SUMMARY:
Randomized, double-blind placebo-controlled phase I trial with the primary aim to investigate safety and tolerability of three ascending dosing schemes of DM-101-PX in birch pollen allergic adults. As an explorative objective, the trial will also investigate the effect of DM-101PX on the allergic symptoms following birch pollen allergen exposure in a chamber. Expanded access to the study treatment is not available.

DETAILED DESCRIPTION:
The study will be carried out in a single study site located in Canada

ELIGIBILITY:
Inclusion Criteria:

* Either sex or any race, aged 18 to 65 years
* Good general health
* A documented clinical history of moderate to severe birch pollen induced allergic rhinitis or rhinoconjunctivitis with symptoms that interfere with daily activities or sleep and remain bothersome despite the use of relevant symptomatic medication, and have been present over at least 2 previous birch pollen seasons
* Birch pollen specific IgE ≥ 0.7 kU/L
* Positive SPT to birch pollen allergen, with wheal diameter ≥ 3 mm
* Body weight ≥ 50 kg and body mass index within the range of 18-35 kg/m2

Exclusion Criteria:

* History or findings on physical examination of any significant disease or disorder which, in the opinion of the Investigator, could put the subject at risk because of participation in the trial, influence the results of the trial or subject's ability to participate in the trial
* Current diagnosis of persistent asthma, or moderate to severe asthma requiring GINA Step 2 or higher treatment, or asthma partially controlled or uncontrolled according to GINA classification in the 6 months before screening
* Significant rhinitis, sinusitis, significant and/or severe allergies not associated with the birch pollen season
* History of asthma deterioration that resulted in emergency treatment or hospitalization in the past 12 months before screening, or a life-threatening asthma attack at any time in the past
* A Forced Expiratory Volume in one second (FEV1) ≤ 75% of predicted value
* History of severe drug allergy, severe angioedema, or systemic allergic reaction of Grade 3 or grater, according to World Allergy Organization (WAO) scale, due to any cause

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | From the first dose to until 14-28 days from the last dose
  Occurrence of treatment emergent adverse events
Adverse Events of Special Interest | From the first dose to until 14-28 days from the last dose
  Occurrence of local injection site reactions and systemic allergic reactions

SECONDARY OUTCOMES:
Subjects Reaching the Maximum Intended Dose | Through the treatment period, an average of 10 weeks
  Number of subjects in each cohort who reach the maximum intended dose

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nilson, Study Director — Desentum Oy; Patricia Couroux, Principal Investigator — Cliantha Research
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to patient level data and related study documents: patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants after Desentum has received marketing authorization from major health authorities (e.g. FDA, EMA), has the legal authority to share the data, and has made the study results publicly available.